CLINICAL TRIAL: NCT06151639
Title: Comparison of The Effects Of General Anesthesia and PECS Block Methods on Blood Leukocyte, Neutrophil, Lymphocyte, and Platelet Counts in Patients With Breast Cancer
Brief Title: Comparison of The Effects Of General Anesthesia and PECS Block Methods on Blood Counts in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Guldeniz Argun, Associate Professor Dr., Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2023-03/130
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: General Anesthesia; PECS block; Neutrophil-Lymphocyte ratio; Platelet-Lymphocyte ratio
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery under general anesthesia: 13 patients were anesthetized intravenous with routine general anesthesia.
  Interventions: Procedure: general anesthesia
- Surgery with Pecs block: 13 patients underwent surgery with PECS block
  Interventions: Procedure: peripheral nerve blocks

INTERVENTIONS:
Procedure: general anesthesia — General anesthesia was performed by muscle relaxant(rocuronium 0,6 mg/kg), opioids(phentanyl 1-2 mcg/kg) and propofol 2mg/kg. Inhation anesthetics and remiphentanyl infusion were used for maintance general anesthesia.
  Groups: Surgery under general anesthesia
Procedure: peripheral nerve blocks — With the help of ultrasonography, at the 2nd rib level, between the fasciae of the pectoralis major and minor muscles at the mid-clavicle level (PECS I block, interpectoral fascial plane block) and at the 4th rib level, at the mid-axillary level, between the fasciae of the pectoralis minor and serratus muscles (PECS II block, pectoroseratal fascial plane block) local anesthesia was applied. In patients who underwent PECS block, a high-frequency linear ultrasonography (Esaote, My LabFive-Genova, Italy) probe and a 50 mm tip insulated needle (echoplex+, Vygon Ecouen-France) were used. 0.200% bupivacaine 15 ml was applied for the PECS I block, and 0.200% bupivacaine 20 ml was applied for the PECS II block, and fascial separation was observed. Sensory control was performed in the breast and axilla area and the patients were taken into surgery.
  Groups: Surgery with Pecs block

SUMMARY:
Regional anesthesia and local anesthetics have proven anti-inflammatory and antitumor effects as well as their analgesic properties.

On this trial, the investigators are searching anesthetic techniques affect on the leukocyte, platelet-lymphocyte count and ratios, total amount of opioids used, and discharge times in patients who will undergo wire localized lumpectomy operation.

DETAILED DESCRIPTION:
For some solid tumors, surgical resection is the best approach available. Surgery causes the release of pro-inflammatory mediators and stimulation of the neuroendocrine system in the perioperative period. Additionally, surgery causes increased sympathetic stimulation and initiates a proinflammatory response to tissue damage. This pro-inflammatory response influences the cell-mediated immune response. Natural killer (NK) cells and CD8+ T cells both have antitumor activities and are associated with cortisol and catecholamine release. It also causes activation of pro-oncogenic cells, regulatory T cells, and type 2 helper T cells. This biological response to surgical stress may result in tumor cell survival and metastasis. Metastatic diseases are the most common cause of death in cancer patients. Exposure to anesthesia during surgery may also play a role in primary relapse or metastatic transformation. Agents used in the induction and maintenance of general anesthesia have interactions with the immune and neuroendocrine systems and may affect the stress response during surgery. Therefore, it is important to choose the best type of anesthesia that will help alleviate sympathetic and/or pro-inflammatory responses while modulating cytokine release and transcription factors/oncogenes. The effect of anesthesia may affect cancer cell survival and ability to metastasize, which can be stimulated not only during surgery but also during the immediate post-operative recovery phase. Studies on the effects of anesthesia methods and anesthetic drugs on tumor recurrence and metastasis are ongoing. It has been shown that volatile anesthetics such as sevoflurane and isoflurane may cause suppression of the immune system by blocking antigen-1-dependent integrin lymphocyte function. Non-volatile anesthetics such as ketamine have been shown to suppress Natural Killer (NK) cell cytotoxicity and inhibit the production of pro-inflammatory cytokines (IL-6 and TNF-α). It has been reported that opioids used alone in pain and pain treatment cause suppression of the immune system through NK activity. Regional anesthesia; It has been hypothesized that it may reduce cancer progression through different mechanisms, including modulation of the sympathetic response, avoidance of the harmful effects of general anesthetics and opioids, and direct immunomodulatory effects of local anesthetics. Peripheral nerve blocks are a regional anesthesia method used to reduce postoperative pain and opioid consumption in many primary tumor resections. In addition to the analgesic properties of local anesthetics and regional anesthesia methods used in regional anesthesia, their anti-inflammatory and antitumor effects have also been proven. The use of ultrasound (US) in peripheral nerve blocks for the last 10 years has increased the success rate in blocks and led to the discovery of new blocks. Fascial plane blocks (FPBs) are regional anesthesia techniques performed by needle insertion and injection into the space between two separate fascial layers. Analgesia is achieved by spreading local anesthetic to the nerves and adjacent tissues moving within this plane. In 2011, Rafael Blanco introduced a new method to analgesia methods after breast surgery by blocking the medial and lateral pectoral nerves of the brachial plexus between the pectoralis major and minor muscles (Pectoral Block I). Pectoral Block II was developed to be effective in axillary interventions. Ultrasound-guided Pectoral Block I and II (PECS I and II) are alternative methods to thoracic epidural and paravertebral blocks in preventing pain after breast surgery. In study, the investigators aimed to compare the effects of general anesthesia and peripheral nerve block (PECS Block) methods on the leukocyte, platelet-lymphocyte count and ratios, the total amount of opioids used, and discharge times in patients who underwent wire localized lumpectomy. It is aimed to ensure that the operation can be performed with peripheral nerve blocks, to protect the patient from immunosuppression that may be caused by general anesthetics and opioids, and to enable early discharge. The originality of the study is to investigate the usability of the PECS Block method not only as a postoperative pain method but also as an anesthesia method during surgery.

In addition, no clinical study has been found in the literature comparing the regional anesthesia method, which is applied only with local anesthetics, with the general anesthesia method.

The study was planned retrospectively. 50 patients who underwent wire localized lumpectomy for breast cancer treatment and diagnosis under general anesthesia (n=25) or PECS block (n=25) were found in hospital records. PECS block was applied to patients who had a high risk of general anesthesia or who did not want to receive general anesthesia during the pandemic. Patients who could not reach a sufficient block level and required additional doses of analgesics were not included in the study. In the PECS I block, local anesthetic was applied between the fascia of the pectoralis major and minor muscles, and in the PECS II block, local anesthetic was applied between the fascia of the pectoralis minor and serratus muscles. The surgery duration, total analgesic amounts pre- and post-operative leukocyte, neutrophil, lymphocyte, platelet levels, and discharge times were evaluated from the records.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral primary breast cancer
* Are decided to undergo wire localized lumpectomy
* Having a risk score of The American Society of Anaesthesiologists (ASA) risk score 1,2 and 3
* Should be over18 years old

Exclusion Criteria:

* Being allergic to the anesthetics
* Opioid or steroid usage before the operation
* Patients who could not reach a sufficient block level and required additional doses of analgesics

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was planned retrospectively. 50 patients who underwent wire localized lumpectomy for breast cancer treatment and diagnosis under general anesthesia (n=25) or PECS block (n=25) were found in hospital records.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
lymphocyte values | postoperative first day
  difference in preoperative and postoperative lymphocyte values between the general anesthesia and PECS block groups
neutrophil values | postoperative first day
  difference in preoperative and postoperative neutrophil values between the general anesthesia and PECS block groups
platelet values | postoperative first day
  difference in preoperative and postoperative platelet values between the general anesthesia and PECS block groups

SECONDARY OUTCOMES:
postoperative Neutrophil/Lymphocyte values | postoperative first day
  diffrence in preoperative and postoperative Neutrophil/Lymphocyte ratios compared to preoperative values between the general anesthesia and PECS block groups
postoperative platelet/lymphocyte ratios | postoperative first day
  difference in preoperative and postoperative platelet/lymphocyte ratios compared to preoperative values between the general anesthesia and PECS block groups
The discharge time | postoperative first day
  The discharge time of patients between the general anesthesia and PECS block groups

OTHER OUTCOMES:
total opioid consumption | intraoperative
  difference between the general anesthesia and PECS block groups

CONTACTS AND LOCATIONS:
Overall Officials: Guldeniz ARGUN, Principal Investigator — Dr. Abdurrahman Yurtaslan Oncology Train and Research Hospita
Locations (1):
- Dr.Abdurrahman Yurtaslan Ankara Oncology Train and Research Hospita, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montejano J, Jevtovic-Todorovic V. Anesthesia and Cancer, Friend or Foe? A Narrative Review. Front Oncol. 2021 Dec 23;11:803266. doi: 10.3389/fonc.2021.803266. eCollection 2021. PMID 35004329
- [Background] Coussens LM, Werb Z. Inflammation and cancer. Nature. 2002 Dec 19-26;420(6917):860-7. doi: 10.1038/nature01322. PMID 12490959
- [Background] Weingart SN, Nelson J, Koethe B, Yaghi O, Dunning S, Feldman A, Kent D, Lipitz-Snyderman A. Association between cancer-specific adverse event triggers and mortality: A validation study. Cancer Med. 2020 Jun;9(12):4447-4459. doi: 10.1002/cam4.3033. Epub 2020 Apr 13. PMID 32285614
- [Background] Forget P, Aguirre JA, Bencic I, Borgeat A, Cama A, Condron C, Eintrei C, Eroles P, Gupta A, Hales TG, Ionescu D, Johnson M, Kabata P, Kirac I, Ma D, Mokini Z, Guerrero Orriach JL, Retsky M, Sandrucci S, Siekmann W, Stefancic L, Votta-Vellis G, Connolly C, Buggy D. How Anesthetic, Analgesic and Other Non-Surgical Techniques During Cancer Surgery Might Affect Postoperative Oncologic Outcomes: A Summary of Current State of Evidence. Cancers (Basel). 2019 Apr 28;11(5):592. doi: 10.3390/cancers11050592. PMID 31035321
- [Background] Deng F, Ouyang M, Wang X, Yao X, Chen Y, Tao T, Sun X, Xu L, Tang J, Zhao L. Differential role of intravenous anesthetics in colorectal cancer progression: implications for clinical application. Oncotarget. 2016 Nov 22;7(47):77087-77095. doi: 10.18632/oncotarget.12800. PMID 27780923
- [Background] Gabriel RA, Swisher MW, Sztain JF, Furnish TJ, Ilfeld BM, Said ET. State of the art opioid-sparing strategies for post-operative pain in adult surgical patients. Expert Opin Pharmacother. 2019 Jun;20(8):949-961. doi: 10.1080/14656566.2019.1583743. Epub 2019 Feb 27. PMID 30810425
- [Background] Bugada D, Lorini LF, Lavand'homme P. Opioid free anesthesia: evidence for short and long-term outcome. Minerva Anestesiol. 2021 Feb;87(2):230-237. doi: 10.23736/S0375-9393.20.14515-2. Epub 2020 Aug 4. PMID 32755088
- [Background] Chong PH, Yeo ZZ. Parenteral Lidocaine for Complex Cancer Pain in the Home or Inpatient Hospice Setting: A Review and Synthesis of the Evidence. J Palliat Med. 2021 Aug;24(8):1154-1160. doi: 10.1089/jpm.2020.0622. Epub 2020 Dec 22. PMID 33351710